CLINICAL TRIAL: NCT05483816
Title: MultiSENSory Stimulation to TArgeT Sensory Loss and ChronIc Pain in NeurOpathic PatieNts
Acronym: SENSATION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ETH Zurich (Other)
Collaborators: Neural Control of Movement laboratory ETH Zurich (Unknown)
Responsible Party: Principal Investigator, Stanisa Raspopovic, Prof. Dr. Stanisa Raspopovic, ETH Zurich
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NeuroengLab
Record Dates: First submitted 2022-07-14; First posted 2022-08-02 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Neuropathy; Neuropathy, Painful; Sensory Neuropathy; Diabetic Neuropathies; Amputation
MeSH Terms: conditions — Neuropathy, Painful; Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Reality and Transcutaneous Electrical Nerve Stimulation (Experimental): for healthy subjects: painful stimulus induction (electrical stimulation) for patients: focus/non focus on pain
  Therapy is released in presence of pain
  Interventions: Combination Product: VR+TENS
- Virtual Reality only (Active Comparator): only VR delivers therapy
  Interventions: Combination Product: VR+TENS

INTERVENTIONS:
Combination Product: VR+TENS — The subjects will receive a therapy that combines electrical pleasant stimulation of the nerves, synchronised with event in virtual reality

SUMMARY:
Neuropathy is a costly and disabling health issue, which consists of a degeneration of the peripheral nerves. Even though the causes may be different, such as diabetes or amputation, the consequences for neuropathic patients are multiple and extremely debilitating. Among the alarming symptoms it implicates, chronic pain and sensory loss are among the most severe ones. Because of the loss of sensations, patients are forced to have an altered gait strategy, an impaired balance and a fivefold increased risk of falling. Furthermore, since they lose sensations and feel numbness in their extremity, they are discouraged in walking, hence leading to a sedentary lifestyle. All of this is worsened by the development of neuropathic pain, which has a high comorbidity with psychological issues, such as depression and anxiety.

Today, proper treatments for neuropathic pain that exclude pharmacological solutions are still missing. This is due to the complexity of the neurobiological mechanisms underlying the origin of neuropathy, the multifaceted physical and psychological nature of pain and the lack of reliable biomarkers.

The aim of this project is to tackle the major problems connected to neuropathy thanks to non-invasive stimulation of the peripheral nervous system. The system is composed of an insole with pressure sensors that captures in real time the force exerted by the subject on the foot and couples this information with parameters of electrical stimulation. Thanks to optimal electrode placement and intensity modulation, subjects are able to perceive in real-time in a somatotopic manner (i.e., under their foot) how they are walking. The aim now is twofold: first the investigators want to couple this stimulation with Virtual Reality (VR) to develop a neuroadaptive non-invasive brain computer interface (BCI) to treat pain and secondly the investigators want to measure through fMRI scans whether the use of the sensory feedback system allows any beneficial plastic changes in the brain. Finally, the investigators want to measure through fMRI scans whether the use of the sensory feedback system allows any beneficial plastic changes in the brain.

DETAILED DESCRIPTION:
One of the notoriously hardest and long-established challenges for the whole scientific community concerns the complete understanding and, consequently, the treatment of neuropathy. This condition results in an altered gait strategy, an impaired balance and a fivefold increased risk of falling. Falling is one of the major health-related problems. In the United Kingdom, more than one fourth of accidents requiring hospital treatment are a consequence of falls. Furthermore, since they lose sensations and feel numbness in their extremity, they are discouraged in walking, hence leading to a sedentary lifestyle (which promotes other long-term complications, e.g. of the cardiovascular system). This has also very severe impacts on the patients' psychological health. Indeed, the comorbidity of neuropathy with anxiety and depression has been estimated to be 59% in the U.S population. Patients may develop neuropathic pain, associable to the aberrant sensory inputs. Experiencing pain impacts even more on gait stability and on the fear of falling. Given the complexity of the underlying mechanisms, chronic neuropathic pain is one of the most prevalent, costly and disabling health issue, hitting a huge portion of the world population. Chronic pain, indeed is estimated to affect approximately 19% of the adult European population. Nowadays, current chronic pain therapies (either behavioural, pharmacological or surgical) are inefficient, as demonstrated by the high prevalence, low rates of functional recovery and the assiduous reliance on opioid analgesics.

The reasons of such lack of efficacy can be attributed to different factors, among which the lack of therapies addressing the multidimensions of pain, as pain is not a unitary phenomenon, rather a multidimensional outcome of sensory-discriminative and motivational-affective components, that should be synergistically accounted for, and the lack of reliable biomarkers: objective indicators of pain are needed to demonstrate therapeutic target engagement, to stratify patients and to predict disease progression or therapeutic responses.

These factors are the main focuses of this study, whose aim is to develop a multisensory platform for pain, detecting pain through physiological recordings and delivering a therapy when such physiological biomarkers are detected. First the detection of pain is exploited through electrophysiology and then the therapy is delivered by means of Virtual Reality (VR) and Transcutaneous Electrical Nerve Stimulation (TENS), in order to target both physiological and affective/cognitive components of neuropathic pain. VR and TENS have already singularly produced encouraging results in literature[26-29]. However, these results are conflicting and not conclusive. The investigators believe that the combination of these technologies, which targets all the different aspects of pain, will really provide a successful and lasting benefit to the patients chronic pain.

Furthermore, the nature of the platform, which includes the use of non-invasive electrical stimulation, allows to recreate sensations in parts of the body where the subjects don't feel sensations anymore. Indeed, thanks to years of research, the Neuro-engineering laboratory found optimal stimulation parameters and electrode placement which are able to elicit sensations far from the electrodes placement. Electrodes are indeed placed on healthy parts of the nerves, but the perceived sensation is in the extremities. This allows to target also another extremely common consequence of neuropathy: sensory loss. This symptom forces patients to have an altered gait strategy, impaired balance and a five-fold increased risk of falling. Therefore, in this study the investigators will monitor also the potential benefits of the platform on these aspects.

As for the imaging sessions, before starting the imaging sessions, patients will be assessed to obtain potential information that might impact on the results.

Healthy participants and patients will be asked to participate in two-three fMRI sessions. Prior to the scanning, a calibration procedure will take place, to understand the subject's stimulation parameters and characterize the location and type of sensations elicited.

During the fMRI sessions, the investigators will examine the neural correlates of the referred perceptions and any pain relief induced using the non-invasive TENS stimulation approach. During these sessions different types of stimulations will be performed (with the TENS stimulation system, with vibrotactile stimulators, and with visual stimulations). Resting state fMRI will be used to examine functional connectivity between different regions of interest. Each fMRI session will last ~70-80 minutes.

ELIGIBILITY:
for healthy:

* Inclusion:

  * Age 18-80
  * Visual acuity>6 on Snellen visual acuity chart
* Exclusion:

  * Pregnancy
  * Cognitive deficits (Mini Mental State Examination<23)
  * Cyber-sickness
  * Prior or current psychological diseases
  * Pacemakers
  * Epilepsy
  * Claustrophobia
  * Other MRI contraindications
  * Unhealed fractures
  * Unhealed wounds
  * Cancerous growth in proximity to feet
  * Swollen, infected or inflamed areas on feet or skin eruptions on feet such as phlebitis, thrombophlebitis or varicose veins

for patients:

* Inclusion:

  * Age 18-80
  * Visual acuity>6 on Snellen visual acuity chart
  * Diagnosis of peripheral neuropathy
  * Pain in lower limbs>=3 cm on VAS scale
* Exclusion:

  * Pregnancy
  * Relevant comorbidities that would affect the outcomes of the study (by judgement of physicians)
  * Ulcers
  * Cognitive deficits (Mini Mental State Examination<23)
  * Cyber-sickness
  * Prior or current psychological diseases
  * Pacemakers
  * Epilepsy
  * Claustrophobia
  * Other MRI contraindications
  * Unhealed fractures
  * Unhealed wounds
  * Cancerous growth in proximity to feet

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in pain level | Through study completion, up to 10 days
  Change in pain level reported by the subjects, 10 cm Visual Analogue Scale (VAS) scale with anchor points 0 = No pain and 10 = Worst imaginable pain, Numerical Pain Rating Scale (NPRS), and the Neuropathic Pain Symptom Inventory (NPSI)
Changes in brain activity and connectivity through functional Magnetic Resonance Imaging (fMRI) before and after the treatment | baseline and 1 week follow-up
  will be measured through functional Magnetic Resonance Imaging (fMRI) sessions
Changes in brain activity and connectivity through functional Magnetic Resonance Imaging (fMRI) between somatotopic and non somatotopic stimulation at feet | baseline, pre-intervention
  The brain activity will be measured while stimulating the subjects in three different locations: 1.somatotopic 2. in-loco 3. at the ankle

SECONDARY OUTCOMES:
Changes in EEG | Through study completion, up to 10 days
  EEG: electroencephalography is a non-invasive measure. A cap is placed on the subject's head and detects the brain activity. In order to do so, a conduction gel (washable with water) is placed on each electrode. We will measure: general Power Spectral Density, frequency bands power (delta, theta, alpha, beta, gamma), connectivity, phase locking value, entropy.
Changes in Skin Conductance signatures | Through study completion, up to 10 days
  Skin Conductance (SC): skin conductance is a measure of the electrodermal activity. It is measured through a couple of non invasive electrodes on the palm of the patient. We will extract features such as peak amplitude, latency, variation, derivative.
Percentage of session completed | post-intervention
  Compliance = % of each session completed.
Changes in Anxiety and Depression | baseline, post-intervention
  measured through validated questionnaires: Beck Anxiety Inventory and Beck Depression inventory
Changes in Quality of life | baseline, post-intervention
  measured through validated questionnaires Neuro-Quality of life
changes in balance | baseline, during the intervention, post-intervention
  Balance will be measured by validated tests (Berg Balance Scale), that range between 0 and 56 (lower values=higher impairment)
changes in the speed to perform the Timed Up and Go (TUG) test | baseline, during the intervention, post-intervention
  Functional mobility will be measured by the Timed Up and Go (TUG) test which measures the time that it takes a person to rise from a chair, walk 7 m, turn around and return and sit in the chair.
changes in the ankle dorsiflexion angle is derived from gait analysis | baseline, during the intervention, post-intervention
  The ankle dorsiflexion angle is derived from gait analysis. The angle of the ankle at the time the foot contacts the floor during a step is derived. This is repeated for at least 5 different walks, and the average of those 5 walks is calculated for further analysis.
changes in speed and cadence in the 10 meter and 6 min walk test | baseline, during the intervention, post-intervention
  In the 10 meter walk test, the time taken by the participant to walk 10 meters is recorded. The test is repeated and the average is taken for analysis.
  In the 6 min walk test, the steps taken by the participant in 6 min walking are recorded.

OTHER OUTCOMES:
Changes in Sensory assessment through Quantitative Sensory Testing (QST) | baseline, during the intervention, post-intervention
  QST: quantitative sensory testing is a set of measurements that measure the sensitivity of subjects. The include: light touch, vibration, hot and cold.
Changes in sensory acuity | baseline, during the intervention, post-intervention
  Sensory discrimination: an object with two extremities distant from 2 to 60 mm are placed on the subject's tested area and the subjects are asked to rate whether they feel 1 or 2 points.
Changes in reflex | baseline, during the intervention, post-intervention
  Reflexes: the ability to have intact reflexes corresponds to healthy nerves. Of particular interest will be the H reflex, where the tibial nerve is stimulated behind the knee and the reflex is measured through electromyography at the calf. We will measure it's latency, amplitude and ratio between M wave and H reflex

CONTACTS AND LOCATIONS:
Overall Officials: Stanisa Raspopovic, Prof. Dr., Principal Investigator — ETH Zurich
Locations (1):
- ETH Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No